CLINICAL TRIAL: NCT05584111
Title: Phase 1 Study to Evaluate the Safety, PK, PD, and Clinical Activity of STC-15, a METTL-3 Inhibitor, in Subjects With Advanced Malignancies
Brief Title: Oral Administration of STC-15 in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: STORM Therapeutics LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STC15-22101
Record Dates: First submitted 2022-09-22; First posted 2022-10-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Cancer
Keywords: Oncology; METTL-3 Inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose Level 1 (Experimental): 30mg capsules, daily administration for 3 week (21 day) cycles
  Interventions: Drug: STC-15
- Dose Level 2 (Experimental): 30mg capsules, MWF administration for 3 week (21 day) cycles
  Interventions: Drug: STC-15
- Dose Level 3 (Experimental): 100mg capsules, MWF administration for 3 week (21 day) cycles
  Interventions: Drug: STC-15
- Dose Level 4 (Experimental): 30mg and 100mg capsules, M-MWF administration for 3 week (21 day) cycles
  Interventions: Drug: STC-15
- Dose Level 5 (Experimental): 30mg and 100mg capsules, M-MWF administration for 3 week (21 day) cycles
  Interventions: Drug: STC-15

INTERVENTIONS:
Drug: STC-15 — STC-15 oral capsules various dosing regimen in 3-week cycles
  Other Names: METTL-3 Inhibitor

SUMMARY:
This Phase 1, multi-center, open-label, first-in-human study evaluates multiple ascending daily oral doses of STC-15 in Q3W treatment cycles in a 3+3 cohort design with dose levels determined by a modified Fibonacci algorithm. The study is designed to systematically assess safety and tolerability, pharmacokinetics, pharmacodynamics and clinical activity of STC-15 in adult subjects with advanced malignancies. Dose levels for further evaluation in expansion cohorts will be selected based on all available PK, pharmacodynamic, target engagement, efficacy, safety, and tolerability data including long-term safety data beyond dose limiting toxicities (DLTs). The study may be amended to evaluate STC-15 in combination with a Food and Drug Administration-approved standard of care treatment regimen, which could encompass targeted/chemotherapy, radiation therapy and/or immunotherapy with immune checkpoint blockers.

ELIGIBILITY:
Key Inclusion Criteria:

* > 18 years of age
* Histologic or cytologic confirmation of advanced malignancy that has failed standard of care (SOC) therapy and no further SOC therapy is available or the subject has declined additional SOC therapy
* Adequate organ and marrow function
* ECOG PS of 0 or 1

Key Exclusion Criteria:

* Treatment with any local or systemic antineoplastic therapy within 3 weeks prior to first dose of STC-15
* Major surgery or radiation within the 3 weeks
* Immune-related AEs from immunotherapy that required permanent discontinuation
* Central nervous system (CNS) disease involvement, or prior history of Grade ≥3 drug-related CNS toxicity.
* Active autoimmune disease that has required systemic treatment in the 2 years prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Screening through end of treatment, approximately 6 months
  To evaluate the incidence, severity, and duration of adverse events
Cmax (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the Cmax concentration over a dosing interval, systemic clearance, volume of distribution at steady-state (Vss), and accumulation ratio from first dose to steady-state.
Tmax (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the time to Cmax (Tmax)
Ctrough (PK) | Screening through end of treatment, approximately 6 months
  To determine observed trough serum concentration (Ctrough)
Terminal elimination half life (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the terminal elimination half-life (t½)
AUC (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine AUC in 1 dosing interval
Average concentration (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the average concentration over a dosing interval
Systemic Clearance (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the systemic clearance
Volume of distribution at steady-state (PK) | Screening through Cycle 2 (each cycle is 21 days)
  To determine the volume of distribution at steady-state (Vss)
Accumulation ratio from first dose to steady-state (PK) | Screening through end of treatment, approximately 6 months
  To determine the accumulation ratio from first dose to steady-state

SECONDARY OUTCOMES:
Efficacy as measured by RECIST 1.1 (DoR) | Screening through disease progression, approximately 6 months
  Determine the duration of response (DoR)
Efficacy as measured by RECIST 1.1 (PFS) | Screening through disease progression, approximately 6 months
  Determine progression-free survival (PFS)/PFS assessed per immune-related response evaluation criteria (iPFS).
Efficacy as measured by RECIST 1.1 (DCR) | Screening through disease progression, approximately 6 months
  Determine the disease control rate (DCR)
Efficacy as measured by RECIST 1.1 (ORR) | Screening through disease progression, approximately 6 months
  Determine the objective response rate (ORR)
Recommended Phase 2 Dose (RP2D) | Screening through 90 days after the last dose of STC-15, approximately 9 months
  determine the RP2D for STC-15

OTHER OUTCOMES:
Assessment of m6A modification of mRNA from peripheral blood | Screening through Cycle 2 (each cycle is 21 days)
  To evaluate the effect of STC-15 on METTL3 enzymatic activity
Assessment of serum cytokines levels | Screening through Cycle 2 (each cycle is 21 days)
  To evaluate immunologic biomarkers in blood and tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Holz, Study Director — STORM Therapeutics
Locations (3):
- United States (3):
  - Honor Health, Scottsdale, Arizona
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No